CLINICAL TRIAL: NCT06753461
Title: Intrahepatic Blood Flow Occlusion Strategies and Postoperative Cardiac Injury Risk in Partial Hepatectomy: a Ten-Year Retrospective Study
Brief Title: Intrahepatic Blood Flow Occlusion and Cardiac Injury Risk in Partial Hepatectomy
Status: Completed | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Principal Investigator, Zhifeng Gao, Associate Professor, Beijing Tsinghua Chang Gung Hospital
Other Study IDs: 24446-4-01
Record Dates: First submitted 2024-12-21; First posted 2024-12-31 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-12

CONDITIONS: Perioperative Myocardial Injury; Myocardial Injury After Non-Cardiac Surgery; Hypotension; Ischemia Reperfusion Injury
MeSH Terms: conditions — Hypotension; Reperfusion Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- No Occlusion: During the entire operation, no blood flow to the liver was occluded.
- Portal Vein Occlusion: During the entire procedure, only the portal vein was occluded.
  Interventions: Procedure: intrahepatic blood flow occlusion
- Pringle Occlusion: Pringle occlusion was performed throughout the operation.
  Interventions: Procedure: intrahepatic blood flow occlusion
- Both Occlusion: Both Pringle occlusion and portal vein block were performed throughout the procedure.
  Interventions: Procedure: intrahepatic blood flow occlusion

INTERVENTIONS:
Procedure: intrahepatic blood flow occlusion — The specified blood vessel is temporarily clamped to achieve the intended blockage of blood flow.
  Groups: Both Occlusion; Portal Vein Occlusion; Pringle Occlusion

SUMMARY:
The goal of this observational study is to examine whether intrahepatic blood flow occlusion strategies during partial hepatectomy are associated with postoperative cardiac injury in patients undergoing hepatectomy. The primary questions it seeks to address are:

1. Are the intrahepatic blood flow occlusion method, the number of occlusions, and the cumulative occlusion time associated with postoperative cardiac injury?
2. How do intrahepatic blood flow occlusion, intraoperative hypotension, and postoperative cardiac injury interact? Participants will contribute their inpatient medical records, including information on medical history, surgical procedures, and anesthesia details.

DETAILED DESCRIPTION:
Liver resection is currently the primary surgical treatment for liver tumors, injuries, and other diseases. With the continuous development of surgical techniques, its application has been expanding. However, intraoperative bleeding and poor surgical field exposure remain major challenges in liver resection, seriously affecting the safety and efficacy of the operation.

Hepatic inflow occlusion is a commonly used technique to address these challenges. It can effectively reduce intraoperative bleeding and improve surgical field exposure. However, it can also lead to hepatic ischemia-reperfusion injury, which may aggravate the damage to the remnant liver and even affect liver regeneration.

Recent studies suggest that hepatic ischemia-reperfusion injury may affect distant organs such as the kidneys, brain, lungs, and heart. However, there is still insufficient clinical evidence, especially regarding myocardial injury. In addition, intraoperative hypotension is a common complication of liver resection and may exacerbate the impact of ischemia-reperfusion injury on the myocardium.

This study intends to construct a model incorporating variables related to intraoperative hepatic ischemia and reperfusion, and analyze the relationship between hepatic inflow occlusion and postoperative myocardial injury in liver resection using logistic regression, while considering the mediating effect of hypotension. The results of this study will provide important clinical evidence for optimizing liver resection strategies, reducing myocardial injury, and improving patient prognosis. This research holds significant scientific and clinical value, and is expected to improve the quality of liver surgery and patient survival rates.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized patients aged ≥18 years who underwent partial hepatectomy between November 28, 2004, and May 20, 2024.

Exclusion Criteria:

1. End-stage renal disease patients (requiring renal replacement therapy)
2. ASA score ≥ 4
3. Lack of intraoperative hepatic portal occlusion data
4. Insufficient perioperative myocardial injury biomarker measurement data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients aged ≥18 years who underwent partial hepatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 2600 (Actual)
Dates: Start 2014-11-28 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Myocardial injury after non-cardiac surgery (MINS) | Within 3 days after sugery
  a high-sensitivity troponin T (hs-TnT) of 20 to <65 ng/L with an absolute change of at least 5 ng/L